CLINICAL TRIAL: NCT01047696
Title: Particulate Air Pollution Exposure and Childhood Acute Respiratory Infections in Guatemala: A Randomized Intervention
Brief Title: Randomised Exposure Study of Pollution Indoors and Respiratory Effects
Acronym: RESPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: World Health Organization (Other); Universidad del Valle, Guatemala (Other); University of Liverpool (Other)
Responsible Party: Prof. Kirk R. Smith, UC Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2003-8-165; R01ES010178 (NIH)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-08

CONDITIONS: Respiratory Tract Infections; Pneumonia
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open fire (No Intervention): Households continuing to use an open fire for cooking and heating
- Chimney stove (Experimental): Households randomized to receive a chimney stove (plancha) for cooking and heating
  Interventions: Device: Plancha

INTERVENTIONS:
Device: Plancha — locally developed chimney stove
  Arms: Chimney stove

SUMMARY:
The purpose of this study was to determine whether reduced exposure to indoor air pollution would reduce ALRI incidence in children <18 months of age. Households were randomized to receive a chimney stove (intervention group) or continue using an open fire for cooking and heating (control group).

DETAILED DESCRIPTION:
Acute lower respiratory infections (ALRI) are the chief killer of children. Most cases are pneumonia and the majority occur among poor children under five years in developing countries. Poverty might be said to be the primary cause, which manifests as malnutrition, including micro-nutrient deficiencies, and lack of access to medical care. Another attribute of poverty is household indoor air pollution (HAP) from use of unprocessed solid fuels such as biomass (wood, animal dung and crop wastes) and coal in simple stoves. A meta-analysis of published observational studies found that young children exposed to smoke from household solid fuel use had a rate of ALRI twice that of children not exposed or where clean fuels were used. Recent studies have shown similar ALRI risks associated with short-term air pollution measurements and other indicators of exposure.

ELIGIBILITY:
Inclusion Criteria:

Households were invited to participate in the study if they met the following inclusion criteria:

* Used only an open fire for cooking and heating
* Had a pregnant woman or child < 4 months residing in the home
* Identified as Mam (the regional ethnic group), and had
* Minimal summer migration (less than 12 weeks per year)

Exclusion Criteria:

Households were excluded from participating if:

* The household was already using a chimney stove for cooking
* There was no child <4 months of age or a pregnant woman residing in the home
* Seasonal migration required the family to move to another region for more than 12 weeks of the year

Max Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 537 (Actual)
Dates: Start 2002-10; Primary Completion 2004-12 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was physician-diagnosed pneumonia in children | Through 18 months of age

SECONDARY OUTCOMES:
Severe (hypoxaemic) and RSV pneumonia | Through 18 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Smith, PhD, MPH, Principal Investigator — UC Berkeley
Locations (1):
- San Lorenzo, Guatemala

REFERENCES:
- [Background] Smith-Sivertsen T, Diaz E, Pope D, Lie RT, Diaz A, McCracken J, Bakke P, Arana B, Smith KR, Bruce N. Effect of reducing indoor air pollution on women's respiratory symptoms and lung function: the RESPIRE Randomized Trial, Guatemala. Am J Epidemiol. 2009 Jul 15;170(2):211-20. doi: 10.1093/aje/kwp100. Epub 2009 May 14. PMID 19443665
- [Background] Diaz E, Bruce N, Pope D, Diaz A, Smith KR, Smith-Sivertsen T. Self-rated health among Mayan women participating in a randomised intervention trial reducing indoor air pollution in Guatemala. BMC Int Health Hum Rights. 2008 Jun 5;8:7. doi: 10.1186/1472-698X-8-7. PMID 18533994
- [Background] Diaz E, Bruce N, Pope D, Lie RT, Diaz A, Arana B, Smith KR, Smith-Sivertsen T. Lung function and symptoms among indigenous Mayan women exposed to high levels of indoor air pollution. Int J Tuberc Lung Dis. 2007 Dec;11(12):1372-9. PMID 18034961
- [Background] McCracken JP, Smith KR, Diaz A, Mittleman MA, Schwartz J. Chimney stove intervention to reduce long-term wood smoke exposure lowers blood pressure among Guatemalan women. Environ Health Perspect. 2007 Jul;115(7):996-1001. doi: 10.1289/ehp.9888. PMID 17637912
- [Background] Diaz E, Smith-Sivertsen T, Pope D, Lie RT, Diaz A, McCracken J, Arana B, Smith KR, Bruce N. Eye discomfort, headache and back pain among Mayan Guatemalan women taking part in a randomised stove intervention trial. J Epidemiol Community Health. 2007 Jan;61(1):74-9. doi: 10.1136/jech.2006.043133. PMID 17183019
- [Result] Smith KR, McCracken JP, Thompson L, Edwards R, Shields KN, Canuz E, Bruce N. Personal child and mother carbon monoxide exposures and kitchen levels: methods and results from a randomized trial of woodfired chimney cookstoves in Guatemala (RESPIRE). J Expo Sci Environ Epidemiol. 2010 Jul;20(5):406-16. doi: 10.1038/jes.2009.30. Epub 2009 Jun 17. PMID 19536077
- [Result] McCracken JP, Schwartz J, Bruce N, Mittleman M, Ryan LM, Smith KR. Combining individual- and group-level exposure information: child carbon monoxide in the Guatemala woodstove randomized control trial. Epidemiology. 2009 Jan;20(1):127-36. doi: 10.1097/EDE.0b013e31818ef327. PMID 19057384
- [Result] Bruce N, Weber M, Arana B, Diaz A, Jenny A, Thompson L, McCracken J, Dherani M, Juarez D, Ordonez S, Klein R, Smith KR. Pneumonia case-finding in the RESPIRE Guatemala indoor air pollution trial: standardizing methods for resource-poor settings. Bull World Health Organ. 2007 Jul;85(7):535-44. doi: 10.2471/blt.06.035832. PMID 17768502